CLINICAL TRIAL: NCT02870738
Title: Comparison of Bladder Directed and Pelvic Floor Therapy in Women With Interstitial Cystitis/Bladder Pain Syndrome
Brief Title: Bladder Directed vs. Pelvic Floor Therapy in IC/BPS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Corewell Health East (Other)
Collaborators: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Kenneth M Peters, MD, Professor and Chairman of Urology, Corewell Health East
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016-253
Record Dates: First submitted 2016-08-12; First posted 2016-08-17 (Estimated); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Cystitis, Interstitial; Painful Bladder Syndrome
MeSH Terms: conditions — Cystitis, Interstitial | interventions — Myofascial Release Therapy; Administration, Intravesical; Lidocaine; Triamcinolone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pelvic Floor Physical Therapy (Active Comparator): One hour of pelvic floor physical therapy twice weekly for 8 weeks
  Interventions: Procedure: Pelvic Floor Physical Therapy
- Bladder Instillations (Active Comparator): Bladder instillation of lidocaine, kenalog, heparin sulphate, and bicarbonate twice weekly for 8 weeks
  Interventions: Drug: Bladder Instillations

INTERVENTIONS:
Procedure: Pelvic Floor Physical Therapy — Internal and/or external myofascial release of the pelvic floor muscles
  Other Names: Myofascial release
  Arms: Pelvic Floor Physical Therapy
Drug: Bladder Instillations — A solution of heparin sulphate 40,000 IU (4 cc of 10,000 units/cc), lidocaine 2% 16 ml, Sodium bicarbonate 8.4% 4 ml and Kenalog 40 mg (1cc) to reach a total fluid volume of 25 ml will be instilled into the bladder with a urinary catheter
  Other Names: xylocaine, triamcinolone
  Arms: Bladder Instillations

SUMMARY:
Women with interstitial cystitis/bladder pain syndrome (IC/BPS) have debilitating urinary frequency and urgency, and chronic pelvic or bladder pain perceived to be related to the bladder. Although many clinicians think that IC/BPS symptoms result from a bladder problem, tight pelvic floor muscles can cause similar symptoms and might be responsible for ICBPS symptoms instead of the bladder. Inadequate assessment of the problem leads to delays in treatment and often years of suffering. This clinical trial will test a bladder directed therapy (bladder instillations) compared to a course of pelvic floor physical therapy (PFPT) to assess the role of the pelvic floor as a major contributor to pelvic pain and voiding dysfunction in adult women with non-ulcerative IC/BPS. Early assessment of the pelvic floor muscles in patients with IC/BPS symptoms may prevent common delays in proper diagnosis and allow for early, more effective treatment.

DETAILED DESCRIPTION:
This will be a prospective randomized trial of pelvic floor therapy vs. bladder directed therapy. The study target population consists of females, aged 18 to 85 years of age with a clinical diagnosis of IC/BPS and symptoms of chronic urinary frequency, pelvic pain/discomfort, and/or urinary urgency. The approximate number of subjects that will be enrolled in the study is 128, 64 women in each treatment group. Women who satisfy all of the eligibility criteria will be enrolled in the study and randomized to receive bladder treatments (instillation of medications into the bladder) or pelvic floor physical therapy.

Outcome measures will include validated questionnaires, voiding diaries, and Global Response Assessment (GRA). The investigators also will evaluate changes in pelvic floor muscle tone and discomfort pre and post treatment, and their relationship to symptom changes. Finally, the investigators will utilize their well-established urine and serum biomarkers evaluations pre and post treatment to determine if they correlate with symptom change.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age 18 to 85 years
* History of patient self-reported of IC/BPS symptoms for at least 6 months.
* Using an approved method of birth control, or surgically sterile, or of non-child bearing age with no menstrual period for the past 12 months
* Must be willing to not start any new medication known to affect bladder or muscle function, and to ideally remain on a stable dose of all other medications through the secondary endpoint.

Exclusion Criteria:

* Active urethral or ureteral calculi, urethral diverticulum, history of pelvic radiation therapy, tuberculous cystitis, bladder cancer, carcinoma in situ (bladder), urethral cancer
* Hunner's lesions found on screening cystoscopy
* Prior investigational or therapeutic bladder instillations for IC/BPS symptoms within the past 3 months
* Lactation, pregnancy, or refusal of medically approved/reliable birth control in women of child-bearing potential.
* Pain, frequency, and/or urgency symptoms only present during menses
* Clinically confirmed urinary tract infection at time of screening
* Participant unable to tolerate insertion of one or two vaginal examining fingers (e.g. Vulvar allodynia)
* Participant had prior course of physical therapy (PT) that included internal (vaginal and/or rectal) manual therapy with connective tissue manipulation by physical therapist for the same symptoms within the past 3 months (prior treatment by therapist with biofeedback, electrical stimulation, or pelvic floor exercises is not exclusionary)
* Participant in the opinion of the investigator has a relevant neurologic disorder that affects bladder and/or neuromuscular function
* Participant has/reports any severe, debilitating or urgent concurrent, medical condition
* Participant has a potentially significant pelvic pathology or abnormality on examination or prior imaging, including prolapse beyond the hymenal ring, pelvic mass, etc., that in the investigators' judgment, could cause or contribute to the clinical symptoms, or require treatment
* Any other condition which, in the investigator's judgment, may increase risk to subject's welfare
* Participation in an investigational trial that uses a study treatment less than 6 months from the date of the screening visit

Note: For the sake of preserving scientific integrity, one or more of the eligibility criteria have been left off the list posted while the trial is ongoing. A full list of eligibility criteria will be posted upon completion of the trial.

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2017-04-21 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Markedly/Moderately Improved on Global Response Assessments | Week 9 (one week after last treatment)
  Proportion of patients in each treatment arm that report Marked or Moderate improvement in symptoms on Global Response Assessments at Week 9 (one week after last treatment)

SECONDARY OUTCOMES:
Change in symptoms | Week 9 (one week after last treatment)
  Change in pelvic floor examination findings and symptoms as measured by questionnaires at Week 9 (one week after last treatment)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth M Peters, MD, Principal Investigator — Corewell Health William Beaumont University Hospital
Locations (1):
- Corewell Health William Beaumont University Hospital, Royal Oak, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Imamura M, Scott NW, Wallace SA, Ogah JA, Ford AA, Dubos YA, Brazzelli M. Interventions for treating people with symptoms of bladder pain syndrome: a network meta-analysis. Cochrane Database Syst Rev. 2020 Jul 30;7(7):CD013325. doi: 10.1002/14651858.CD013325.pub2. PMID 32734597